CLINICAL TRIAL: NCT03651102
Title: Efficacy and Safety of Low Dose Thalidomide in Transfusion Dependent Thalassemia Patients of Pakistan
Brief Title: Efficacy and Safety of Low Dose Thalidomide in Transfusion Dependent Thalassemia
Acronym: Thal-Thalido
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Blood Diseases Clinic (Other)
Collaborators: University of Peshawar (Other)
Responsible Party: Principal Investigator, Muhammad Tariq Masood Khan, Consultant Haematologist; Research Associate, Blood Diseases Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDT
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Thalassemia
Keywords: Thalidomide; Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Thalidomide; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thalidomide in combination with hydroxyurea (Experimental): All the study patients refractory to hydroxyurea will be given thalidomide at an average dose of 2mg/kg/day (range 1-4mg/kg/day). Participants will also be continued on hydroxyurea at a dose of 10-20 mg/kg/day.
  Interventions: Drug: Thalidomide and Hydroxyurea

INTERVENTIONS:
Drug: Thalidomide and Hydroxyurea — Dosage: Thalidomide 1-4mg/kg/day, Hydroxyurea 10-20mg/kg/day

SUMMARY:
Thalidomide is known to have hypnosedative, immuno-modulatory and anti-angiogenic effects. The drug is widely used in several neoplastic disorders (e.g. multiple myeloma and malignant melanoma), inflammatory conditions (e.g. Crohn's disease) and skin disorders (e.g. leprosy). Thalidomide has been successfully used in adult thalassemia patients. The current study explores its role in transfusion-dependent thalassemia patients.

ELIGIBILITY:
Inclusion Criteria:

* Transfusion dependent thalassemia patients refractory to Hydroxyurea

Exclusion Criteria:

* Those with active systemic comorbidity, with past personal or family history of thrombophilia, recent fracture or recent major surgery

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Haemoglobin Level | 6-24 months
  mg/dL
Response Rate (Excellent, Good, Partial and No response) | 6-24 months
Adverse Effects | 6-24 months

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tariq M Khan, MBBS, PhD, Principal Investigator — Blood Diseases Clinic; Zahid Ali, PharmD, MPhil, Study Director — Department of Pharmacy, University of Peshawar
Locations (1):
- Blood Diseases Clinic, Peshawar, Khyber Pakhtukhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Ren Q, Zhou Y, Li P, Lin W, Yin X. Thalidomide has a significant effect in patients with thalassemia intermedia. Hematology. 2018 Jan;23(1):50-54. doi: 10.1080/10245332.2017.1354427. Epub 2017 Jul 18. PMID 28718348
- [Background] Ren Q, Zhou YL, Wang L, Chen YS, Ma YN, Li PP, Yin XL. Clinical trial on the effects of thalidomide on hemoglobin synthesis in patients with moderate thalassemia intermedia. Ann Hematol. 2018 Oct;97(10):1933-1939. doi: 10.1007/s00277-018-3395-5. Epub 2018 Jun 22. PMID 29931453
- [Background] Masera N, Tavecchia L, Capra M, Cazzaniga G, Vimercati C, Pozzi L, Biondi A, Masera G. Optimal response to thalidomide in a patient with thalassaemia major resistant to conventional therapy. Blood Transfus. 2010 Jan;8(1):63-5. doi: 10.2450/2009.0102-09. No abstract available. PMID 20104280
- [Background] Ricchi P, Costantini S, Spasiano A, De Dominicis G, Di Matola T, Cinque P, Ammirabile M, Marsella M, Filosa A. The long-term and extensive efficacy of low dose thalidomide in a case of an untransfusable patient with Non-Transfusion-Dependent Thalassemia. Blood Cells Mol Dis. 2016 Mar;57:97-9. doi: 10.1016/j.bcmd.2016.01.003. Epub 2016 Jan 16. PMID 26810455
- [Background] Aguilar-Lopez LB, Delgado-Lamas JL, Rubio-Jurado B, Perea FJ, Ibarra B. Thalidomide therapy in a patient with thalassemia major. Blood Cells Mol Dis. 2008 Jul-Aug;41(1):136-7. doi: 10.1016/j.bcmd.2008.03.001. Epub 2008 Apr 24. No abstract available. PMID 18439858
- [Background] Chen J, Zhu W, Cai N, Bu S, Li J, Huang L. Thalidomide induces haematologic responses in patients with beta-thalassaemia. Eur J Haematol. 2017 Nov;99(5):437-441. doi: 10.1111/ejh.12955. Epub 2017 Sep 27. PMID 28850716
- [Background] Fard AD, Hosseini SA, Shahjahani M, Salari F, Jaseb K. Evaluation of Novel Fetal Hemoglobin Inducer Drugs in Treatment of beta-Hemoglobinopathy Disorders. Int J Hematol Oncol Stem Cell Res. 2013;7(3):47-54. PMID 24505535
- [Background] Gambari R. Foetal haemoglobin inducers and thalassaemia: novel achievements. Blood Transfus. 2010 Jan;8(1):5-7. doi: 10.2450/2009.0137-09. No abstract available. PMID 20104272
- [Derived] Ali Z, Ismail M, Rehman IU, Rani GF, Ali M, Khan MTM. Long-term clinical efficacy and safety of thalidomide in patients with transfusion-dependent beta-thalassemia: results from Thal-Thalido study. Sci Rep. 2023 Aug 21;13(1):13592. doi: 10.1038/s41598-023-40849-4. PMID 37604857